CLINICAL TRIAL: NCT01978210
Title: Development of a Manualized Wireless Moisture Pager Intervention for Teaching Toileting in Children With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Autism Treatment Network (Network)
Responsible Party: Principal Investigator, Daniel Mruzek, Associate Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Moisture Pager Intervention
Record Dates: First submitted 2013-10-24; First posted 2013-11-07 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Autism; Enuresis; Incontinence
Keywords: autism; enuresis; toilet-training
MeSH Terms: conditions — Autistic Disorder; Enuresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wireless Moisture Pager (Experimental): Parent(s) of subjects will participate in training and follow-up sessions in a manualized toilet training intervention for their child that incorporates use of a wireless moisture pager.
  Interventions: Device: Wireless Moisture Pager (WMP)
- Standard Behavioral Treatment (Active Comparator): Parent(s) of subjects will participate in training and follow-up sessions in a toilet training intervention for their child that incorporates use of the Autism Treatment Network's Toilet Training Tool Kit. The Tool Kit is a publication widely available to parents and clinicians that is designed to serve as an aid in the toilet training of children with autism. In this study, it is being used as a standard treatment control.
  Interventions: Device: Wireless Moisture Pager (WMP)

INTERVENTIONS:
Device: Wireless Moisture Pager (WMP) — The WMP is composed of a three key components: (1) the disposable sensor; (2) the transmitter; and (3) the receiver. The disposable sensor is placed by the parent in the child's underwear and detects small amounts of urine. The transmitter is housed in hardened plastic, attached to the disposable sensor, and, upon activation, emits a radio signal to the receiver. The receiver is an iPod-based app that emits an audible and/or vibration signal to the parent and child at the onset of a toileting accident. A step-by-step manualized curriculum is used to teach parents how to incorporate the device in the toilet training of their child.

SUMMARY:
This pilot study is designed to investigate the feasibility of comparing a standard behavioral intervention and an innovative intervention that incorporates the use of a wireless moisture alarm in training children with autism how to independently use the toilet for urination. We hypothesize that the study protocol will be feasible, as measured through review of achieved recruitment targets, successful randomization, and >80% retention of subjects with com- plete data collection. Our second hypothesis is that therapists will deliver experimental and standard behavioral treatment intervention with ≥80% fidelity and parents in both intervention groups will adhere to the intervention with ≥80% fidelity. A secondary aim of this study is to examine trends in outcome data by conducting a small RCT (N = 30) of wireless moisture alarm and standard behavioral toilet training, with the hypothesis that the moisture alarm intervention will result in fewer toileting accidents, a higher rate of toileting success and greater parental satisfaction.

ELIGIBILITY:
Inclusion Criteria:

1. Age 3-6 years old
2. ASD diagnosis confirmed by licensed professional through administration of the ADOS or ADOS-2, depending upon availability of data
3. Status consistent with DSM-IV (or DSM-V, depending upon availability) diagnostic criteria for primary daytime enuresis (with exception of criterion that child is at least 5 years old), confirmed by the K- SADS
4. A positive determination of readiness for toilet training, as determined through aToileting Readiness Checklist developed through a review of relevant literature on toilet training with children with autism (with 4 or more of 7 signs in the checklist, with 3 of these criteria required).
5. Consent from parent

Exclusion Criteria:

1. Medical conditions that would interfere with toilet training procedures (e.g., physical disabilities)
2. Physical disorder that may contribute to incontinence (e.g., diabetes, urinary tract infection, or seizures)
3. Anticipation of medication changes to occur during the 3-month intervention period
4. Medication for enuresis
5. A parent report that the child has urinated into a toilet 2 times or more when toilet trips are initiated by child, AND/OR 20% or more of the total instances in which a caretaker had initiated a toileting opportunity (to be estimated by study team member during initial conversation. If parent is unsure, they may be asked to monitor toileting behavior for a week, and the team member can call back to review with parent).
6. Parent report that the child has participated in systematic training efforts, under the guidance of a clinician (e.g., physician, psychologist) for more than 8 weeks (total) in the previous 6months.
7. Active drug or alcohol use or dependence on the part of the parent that, in the opinion of the site investigator, would interfere with adherence to study re- quirements.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2013-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Total number of participants successfully recruited | 3-month intervention
  As a pilot study, a key outcome variable is the number of families successfully recruited for participation in this study involving intensive toilet training administered by parents.
Percentage of participants retained across the life of the study | 3 months
  80% retention across the life of the study will be considered evidence of satisfactory retention of participating families.
Treatment Fidelity (Interventionists) | 3 months
  Digitally recorded 2-hour initial parent training sessions will be scored by independent raters using an intervention fidelity checklist to assess the degree to which interventionists are successful in delivering the treatments. Scores of 80% fidelity will be considered evidence of satisfactory treatment fidelity.
Fidelity of Parent Implementation | 3 Months
  Using fidelity checklists, interventionists will rate parents' participation in toilet training intervention, as well as their fidelity to the key components of the intervention.

SECONDARY OUTCOMES:
Rate of toileting accidents | 6 months
  Data logs maintained by parents during the 3 consecutive days prior to office visits will be used to measure toileting accidents. These data will be used to test the hypothesis that the WMP group will have fewer toileting accidents than the SBT group.This will be assessed at 3 months (close of active intervention) and at a 6-month follow-up appointment.
Participants' Daily Rate of Toilet Use for Urination | 6 months
  Toileting logs maintained by parents for 3 consecutive days prior to study visit will be used to measure the daily rate of toilet use for participants. These data will be used to test the hypothesis that children in the WMP group will demonstrate more rapid acquisition of toileting skills than children in the SBT group. This will be assessed at 3 months (close of active intervention) and at a 6-month follow-up appointment.
Parent Satisfaction with Toilet Training Intervention | 6 months
  A parent satisfaction rating scale will be used to measure their satisfaction with their experience with the toilet training intervention for their child. These data will be used to test the hypothesis that parents participating in the WMP intervention will report overall greater satisfaction with their training experience relative to the SBT group. This will be assessed at 3 months (close of active intervention) and at a 6-month follow-up appointment.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel W Mruzek, PhD, Principal Investigator — University of Rochester
Locations (3):
- United States (3):
  - University of Rochester Medical Center, Rochester, New York
  - Nationwide Children's Hospital, Columbus, Ohio
  - Whitney Loring, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Investigators can contact the responsible party to obtain de-identified data.

REFERENCES:
- [Derived] Mruzek DW, McAleavey S, Loring WA, Butter E, Smith T, McDonnell E, Levato L, Aponte C, Travis RP, Aiello RE, Taylor CM, Wilkins JW, Corbett-Dick P, Finkelstein DM, York AM, Zanibbi K. A pilot investigation of an iOS-based app for toilet training children with autism spectrum disorder. Autism. 2019 Feb;23(2):359-370. doi: 10.1177/1362361317741741. Epub 2017 Dec 7. PMID 29212345